CLINICAL TRIAL: NCT05135988
Title: Caring for Children in Vital Distress: Assessment of Paramedical Uses and Benefits of a Software
Brief Title: Caring for Children in Vital Distress
Acronym: EasyPedia
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/581
Record Dates: First submitted 2021-10-25; First posted 2021-11-26 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Emergencies; Children
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children in vital distress
- Health care givers: Experts in vital distress care Non experts in vital distress care

SUMMARY:
Errors during a stressful pediatric critical situation occur more frequently than thought. The main aim of the study is to quantify the number and the type of errors made by pediatric paramedical teams during the management of vital emergencies (medication dosage calculation, compliance with algorithms for management of cardiac arrest…). Then, simulations with and without the EasyPédia software will be compared during a high-fidelity simulation of a standardized pediatric cardiac arrest scenario in order to evaluate its impact on reducing errors during the management of a resuscitation.

This study will be a single-center and observational trial in the pediatric intensive care unit of the Besançon University Hospital.

DETAILED DESCRIPTION:
The study is divided in two parts :

Part 1 : non-interventional study Part with children in vital distress enrollment. Fifteen patients will be recruited over a period of 1 year in the intensive care unit.

Part 2 : high-fidelity simulation tests

Part at a simulation platform with assessment of the EasyPedia software. Sixty health care givers divided in 2 groups, experts (intensive care units and specialist mobile emergency units) and non experts (pediatric medicine and pediatric emergencies units) in vital distress care, will be included over a period of 4 months. They will be submitted to two simulation scenarios : with and without the EasyPedia software.

The first part follows a case-only observational study model and the second part follows a case-crossover one.

Concerning the time perspective, the first part is a cross-sectional study and the second part is prospective.

ELIGIBILITY:
Part 1 in intensive care unit :

Inclusion Criteria:

* Patients in vital distress taken in charge in intensive care unit : transported by the specialist mobile emergency units, transferred from an other unit of the Besancon University Hospital or from a peripheral hospital on medical decision
* Children from 0 to 15 years

Exclusion Criteria:

* Premature newborns and patients transported by the specialist mobile emergency units or transferred from an other unit of the Besancon University Hospital on medical decision not presenting a vital emergency following evaluation of the medical team of the intensive care unit
* Subject being in the period of exclusion from another study or provided by the national volunteer file

Part 2 in simulation :

Inclusion criteria

- Expert teams of doctor and paramedics (10 from pediatric intensive care unit and specialist mobile emergency units) and non expert teams of doctor and paramedics (10 from pediatric medicine and pediatric emergencies units)

Exclusion criteria

* Non-consenting doctor or paramedic
* Doctor or paramedic who has worked at night for less than 48 hours
* Care givers under guardianship ou curatorship

Ages: 0 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Part 1 : children in vital distress taken in charge in the Besancon University Hospital Part 2 : health care givers from the Besançon University Hospital
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of the practices of paramedical teams in the care of children in vital distress | Day 0
  Quantification of the number and type of errors made by pediatric paramedical teams during vital emergency management (medication dosage calculation, compliance with algorithms for management of cardiac arrests…), in part 1 of the study

SECONDARY OUTCOMES:
Evaluation of the EasyPedia software impact on reducing the number of errors | Month 4
  Quantification of error-reduction numbers using EasyPedia in high-fidelity simulation, in part 2 of the study
Evaluation of non-technical skills within a team | Month 4
  Evaluation of non-technical skills within a team (communication, coordination, TEAM-score…) in part 2 of the study
Evaluation of the EasyPedia software impact on the anxiety of the medical team members during a simulated critical situation measured with visual analogue scale | Month 4
  Evaluation of the medical team member's anxiety in part 2 of the study using a visual analogue scale [VAS] ranging from 0 (not anxious at all) to 10 (very anxious), before and after the simulation session.
Evaluation of the EasyPedia software impact on the anxiety of the medical team members during a simulated critical situation measured with Strate Trait Anxiety Inventory | Month 4
  Evaluation of the medical team member's anxiety in part 2 of the study using the Strate Trait Anxiety Inventory (STAI Y1/Y2) ranging from 20 (low anxiety) to 80 (high anxiety) for each form, before and after the simulation session.
Evaluation of the EasyPedia software impact on the stress of the medical team members during a simulated critical situation measured with cortisol level | Month 4
  Evaluation of the medical team member's stress in part 2 of the study using measurement of salivary cortisol levels (in nM/L), before and after (juste after and 15 min later) the simulation session.
Evaluation of the EasyPedia software impact on the stress of the medical team members during a simulated critical situation measured with heart rate | Month 4
  Evaluation of the medical team member's stress in part 2 of the study using measurement of heart rate variability using a heart rate monitor belt throughout the simulation session.
Evaluation of the medical team member self-efficacy during a simulated critical situation | Month 4
  Evaluation of self-efficacy perception after the session using a visual analogue scale [VAS] ranging from 0 (totally unable) to 10 (fully capable), in part 2 of the study
Evaluation of the EasyPedia software usability | Month 4
  Evaluation of the EasyPedia software usability using a User Experience Questionnaire (UEQ) with 6 scales (attractiveness, perspicuity, efficiency, dependability, stimulation, novelty) divided into 26 items, after the simulation session with the software, in part 2 of the study. The range of the scales is between -3 (horribly bad) and +3 (extremely good).

CONTACTS AND LOCATIONS:
Locations (1):
- Besançon University Hospital, Besançon, Not in US/Canada, France